CLINICAL TRIAL: NCT04481958
Title: Implementation of Injury Prevention Training and an Associated Implementation Strategy in Youth Handball: A Pilot Study of the I-PROTECT Model
Brief Title: Implementation of the I-PROTECT Model
Acronym: I-PROTECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid-19 restrictions, handball training was only performed about 2 months at the start of the season, and intervention and evaluation could not be conducted as planned.
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Eva Ageberg, PhD, Professor, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014/713
Record Dates: First submitted 2020-07-08; First posted 2020-07-22 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Athletic Injuries
Keywords: Physical activity; Preventive therapy; Adolescent; Health plan implementation; Behaviour change
MeSH Terms: conditions — Athletic Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single case study, purposeful sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- I-PROTECT model (Experimental): The I-PROTECT model is an end-user-driven intervention including evidence-based, theory-informed, and context-specific injury prevention training for youth handball, and an associated implementation strategy.
  Interventions: Behavioral: I-PROTECT

INTERVENTIONS:
Behavioral: I-PROTECT — The I-PROTECT model is based on existing research and knowledge of experts in sport medicine, sport psychology and implementation science, with the involvement of end-users throughout the process. The interdisciplinary intervention includes exercises based on physical and psychological principles of effective injury prevention training, specifically tailored for youth handball players, and support for developing a continuous implementation strategy. The intervention is delivered through a mobile application (the I-PROTECT GO), including modules tailored for coaches, players, club administrators, and caregivers, respectively. Coaches are introduced to the intervention in a workshop, and they will conduct the exercises with their teams during handball practice. Due to pandemic restrictions, the mobile application could not be finalized, and only the module for coaches was available.

SUMMARY:
Evidence-based injury prevention training is highly effective in reducing sport-related musculoskeletal injuries in youth. However, this training has so far had limited public health impact because it is not widely or properly implemented or sustained. In this single case study with youth teams from two handball clubs in Southern Sweden, the aim is to test the I-PROTECT model, featuring injury prevention training and an associated implementation plan. The main hypothesis is that the intervention will result in higher motivational and volitional levels in relation to injury prevention training.

DETAILED DESCRIPTION:
This is a pilot study included in the "Implementing injury Prevention training ROutines in TEams and Clubs in youth Team handball (I-PROTECT)" project (Ageberg et al, 2019, 2020). The overall aim of I-PROTECT is to achieve wide-spread, sustained and high-fidelity use of evidence-based injury prevention training in youth handball through behavior change at multiple levels within the sports delivery system (individual and organizational levels). The I-PROTECT model is evidence-based, theory-informed, and context-specific injury prevention training specifically tailored for youth handball players, incorporating physical and psychological components and an associated implementation strategy. The process of developing the I-PROTECT model has been described (Ageberg et al 2020). The current study is a prospective single case study for initial testing and evaluation of the I-PROTECT model (i.e., before the model is implemented in a larger scale study). The reporting will adhere to the SCRIBE guidelines. All youth teams in the two clubs with representatives of the stakeholder group overseeing the I-PROTECT project will use the I-PROTECT model for one handball season. The Health Action Process Approach (HAPA) theory will be used to evaluate behavior change among players, coaches and club administrators. The Reach, Effectiveness, Adoption, Implementation, and Maintenance Sport Setting Matrix (RE-AIM SSM) framework will be used to guide the evaluation of implementation outcomes of the I-PROTECT model among all stakeholders (players, coaches, club administrators, caregivers).

The main hypothesis is that the intervention increases scores in HAPA questions in coaches from pre- to post intervention by at least 30%, indicating higher motivational and volitional levels in relation to injury prevention training post intervention (end of season) compared to pre-intervention (baseline). A preliminary sample size calculation indicates that 42 coaches are needed to detect a clinically relevant change in behavior of at least 30% (baseline vs post intervention) with 80% power at the 5% significance level. Secondary outcomes will be: i) HAPA questions among players and club administrators; ii) RE-AIM SSM questions, descriptive data, and/or mobile application data among all stakeholders (players, coaches, club administrators, caregivers). Interviews (e.g., focus groups) with end-users will be conducted to enable an in-depth understanding of the feasibility, acceptability and usability of the program, including its packaging. An "exit strategy" will be employed to refine the model, address any potential barriers for implementation and sustainability, and embed the I-PROTECT model into the organizations that have participated in the study.

Due to pandemic restrictions, handball training was only performed as usual about 2 months at the start of the season, and evaluation of the I-PROTECT-model could not be conducted as planned. Nineteen teams with their coaches, players, and caregivers included (approx. 700 participants in total). The following data was collected:

* Main outcome: HAPA questions for coaches at baseline and at end-of-season
* Secondary outcomes: HAPA and RE-AIM questions caregivers at baseline

ELIGIBILITY:
Stakeholders (players, coaches, caregivers, club administrators) of all youth teams (13-17 years) in two community handball clubs will be eligible for participation.

Inclusion Criteria:

* Players: ages 13-17 years and training ≥2 times/week in a team
* Coaches: leading ≥1 training session/week
* Caregivers: directly associated with the eligible players
* Club administrators: engagement in the issues of sports injury, coach education - or policy development for youth players

Exclusion Criteria

* Employed/paid players
* Stakeholder other than the groups listed in inclusion criteria

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Health Action Process Approach questions for coaches | Baseline to end-of-season (after approx. 8 months)
  An adapted version of the Health Action Process Approach (HAPA), specifically related to injury prevention training for youth team handball, has been developed and adapted for coaches. The questions focus on motivational strategies (e.g., risk perception, outcome expectancies) and volitional strategies (e.g., action planning, maintenance self-efficacy) for behavior change regarding injury-prevention training.

SECONDARY OUTCOMES:
Descriptive information about the Covid-19 pandemic and use of I-PROTECT (coaches) | Baseline to end-of-season (after approx. 8 months)
  Questions to coaches about use of I-PROTECT before and during pandemic restrictions
Health Action Process Approach and Reach, Effectiveness, Adoption, Implementation, and Maintenance Sport Setting Matrix questions among caregivers | Baseline
  Health Action Process Approach (HAPA) and Reach, Effectiveness, Adoption, Implementation, and Maintenance Sport Setting Matrix (RE-AIM SSM), specifically related to injury prevention training for youth team handball, adapted for caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PhD, Principal Investigator — Department of Health Sciences, Lund University, Lund, Sweden
Locations (1):
- Eva Ageberg, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Share published data on reasonable request.

REFERENCES:
- [Background] Ageberg E, Bunke S, Nilsen P, Donaldson A. Planning injury prevention training for youth handball players: application of the generalisable six-step intervention development process. Inj Prev. 2020 Apr;26(2):164-169. doi: 10.1136/injuryprev-2019-043468. Epub 2020 Feb 4. PMID 32019772
- [Background] Ageberg E, Bunke S, Lucander K, Nilsen P, Donaldson A. Facilitators to support the implementation of injury prevention training in youth handball: A concept mapping approach. Scand J Med Sci Sports. 2019 Feb;29(2):275-285. doi: 10.1111/sms.13323. Epub 2018 Nov 8. PMID 30339309